CLINICAL TRIAL: NCT05805072
Title: An Open Label, Single Arm, Single-Center Exploratory Study to Evaluate the Efficacy and Safety of Selinexor and HAAG +/- HMA in Relapsed/Refractory Acute Leukemia (AML) Patients
Brief Title: Selinexor and HAAG With/Without HMA in Relapsed/Refractory Acute Leukemia (AML) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Selinexor+HAAG+HMA
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Relapsed/Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — selinexor; Homoharringtonine; Cytarabine; aclacinomycins; Granulocyte Colony-Stimulating Factor; Decitabine; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Selinexor+HAAG±HMA (Experimental)
  Interventions: Drug: Selinexor; Drug: Homoharringtonine; Drug: Cytarabine; Drug: Aclacinomycin; Drug: Granulocyte Colony-Stimulating Factor; Drug: Decitabine; Drug: Azacitidine

INTERVENTIONS:
Drug: Selinexor — Selinexor 60 mg/day, orally on d1,4,8,11
Drug: Homoharringtonine — Homoharringtonine 1 mg/day intravenously on days 3 to 9
Drug: Cytarabine — cytarabine 10 mg/m2 q12h, intravenously on days 3 to 9
Drug: Aclacinomycin — aclacinomycin 10 mg/day intravenously on days 3 to 6
Drug: Granulocyte Colony-Stimulating Factor — granulocyte colony-stimulating factor 50-600 mcg/m2/day intravenously from days 2 to start, this dosage will be adjusted according to the hemogram,
Drug: Decitabine — Decitabine 20 mg/m2/day intravenously on days 1 to 5.
Drug: Azacitidine — Azacitidine 20 mg/m2/day subcutaneously on days 1 to 7

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of selinexor and HAAG +/- HMA in relapsed/refractory acute leukemia (AML) patients.

DETAILED DESCRIPTION:
This protocol corresponds to a single-center, open-label, single-arm, exploratory study designed to determine the efficacy and safety of the combination of selinexor with HAAG +/- HMA in patients with relapsed or refractory AML. The patients who respond to this combination treatment will undergo allogeneic hematopoietic stem cell transplantation and post-transplantation maintenance treatment according to patient's wishes.

Each cycle of treatment will compromise 2 weeks of selinexor treatment, and at least two weeks off treatment. The new cycle will not start if there is an ongoing grade 3 or higher non-hematologic toxicity or persistent grade 3 neutropenia in patients achieving CR.

Study design allows 20 patients. Treatment will consist of selinexor 60 mg/day orally on d1,4,8,11, HHT 1 mg/day intravenously on days 3 to 9, cytarabine 10 mg/m2 q12h, intravenously on days 3 to 9, aclacinomycin 10 mg/day intravenously on days 3 to 6, G-CSF 50-600 mcg/m2/day intravenously from days 2 to start, this dosage will be adjusted according to the hemogram, DAC 20 mg/m2/day intravenously on days 1 to 5. Whether to add hypomethylating agents was decided by the investigator according to the patient's disease degree and tolerance status. If patients had previously been exposed to decitabine, azacitidine will added this regimen, AZA 20 mg/m2/day subcutaneously on days 1 to 7.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥18 years.
2. Diagnosis of AML (defined according to the 5th of the World Health Organization [WHO] 2022 criteria) of any type except for acute promyelocytic leukemia (APL; AML M3)and the following conditions were met: Relapsing or refractory AML
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
4. Female patients of child-bearing potential must have a negative serum pregnancy test at screening and agree to use two reliable methods of contraception for six months after their last dose of medication.
5. Patients whose expecting survival time will be more than 3 months.
6. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.

Exclusion Criteria:

1. AML transformed from chronic myeloid leukemia.
2. Patients with APL/AML M3.
3. Presence of CNS leukemia.
4. Uncontrolled infection or other serious disease.
5. Unstable cardiovascular function: Cardiac ejection fraction (EF)<0.5, or congestive heart failure (CHF) of NYHA Class ≥ 2.
6. Unstable Liver and kidney function:TBLL≥2.0 mg/dl, AST≥3×ULN, Ccr≥50 ml/min, SpO2<92%.
7. Known human immunodeficiency virus (HIV) infection.
8. Active hepatitis B or hepatitis C infection.
9. Pregnant and lactating women. Patients with other commodities that the investigators considered not suitable for the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With CR/CRi | End of cycle 1 and 2 (each cycle is 28 days)
  Number of Participants With CR/CRi
  CR: Absolute Neutrophil count (ANC) >1.0x10^9/L, Platelet count >100x10^9/L, Bone marrow blasts <5%, no Auer rods, no evidence of extramedullary disease.
  CRi: Same as CR, but ANC may be <1.0x10^9/L and/or Platelet count <100x10^9/L

SECONDARY OUTCOMES:
Number of Participants With ORR | End of cycle 1 and 2 (each cycle is 28 days)
  ORR =CR+CRi+PR+MLFS
  PR: Absolute Neutrophil count (ANC) >1.0x10^9/L, Platelet count >100x10^9/L, at least a 50% decrease in the percentage of marrow aspirate blasts to 5-25%, or marrow blasts <5% with persistent Auer rods.
  MLFS: Bone marrow blasts <5%, no Auer rods, no evidence of extramedullary disease
Percentage of Patients Transplanted After Induction Therapy (Stem Cell Transplantation) | 1-2 induction cycles (4 - 8 weeks)
  Rate of ASCT: Percentage of patients being transplanted after induction therapy (stem cell transplantation)
Progression-Free Survival | Time from registration to event, max 2 years
  Progression-free survival (PFS): was calculated from the time of informed consent to the date of recurrence or death, whichever occurred first. Patients were censored at the date of the last follow-up visit if they were alive without relapse.
  Disease progression was defined as presence of >50% increase in bone marrow blasts to a level of at least 50% and/or a doubling of the percentage of peripheral blood blasts to a level of at least 50%.
Overall Survival | Time from registration to event, max 2 years
  Overall survival (OS) was calculated from the date of informed consent to the date of death. Patients still alive at the end of follow-up were censored at the last date of follow-up.
Number of adverse events | End of cycle 1 and 2 (each cycle is 28 days)
  Adverse events are evaluated with CTCAE V5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No